CLINICAL TRIAL: NCT06163391
Title: A Multicenter, Open-label, Phase 1 Study to Evaluate the Safety and Preliminary Efficacy of SOT201 in Patients With Advanced/Metastatic Solid Tumors
Brief Title: A Study to Assess Safety and Efficacy of SOT201 in Patients With Advanced/Metastatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SOTIO Biotech AG (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC201; VICTORIA-01 (Other: SOTIO Biotech AG); 2023-504330-21-00 (Other: EU CT number)
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: Checkpoint inhibition plus RLI-15; SOT201; SC201; VICTORIA-01; RLI-15/CPI fusion protein; Immunocytokine
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: 6 cohorts, multiple-dose escalation, Bayesian optimal interval design (BOIN) trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SOT201 (Experimental): SOT201 will be administered intravenously once every 21 days
  Interventions: Drug: SOT201

INTERVENTIONS:
Drug: SOT201 — intravenous infusion

SUMMARY:
This is a Phase 1, open-label, dose escalation study to assess the safety, tolerability, and preliminary efficacy of SOT201 as monotherapy for participants aged 18 years or above with advanced unresectable or metastatic solid tumors

During dose escalation, the recommended dose(s) of SOT201 given every 3 weeks (Q3W) will be determined

DETAILED DESCRIPTION:
Duration of the study for a participant will include:

Screening period: Up to 21 days before day 1 of cycle 1 (can be prolonged up to 42 days, if required due to fresh biopsy) Treatment Period: enrolled and exposed participants will receive continuous treatment until progressive disease (PD), or an occurrence of an unacceptable AE, a withdrawal of consent, or until other permanent discontinuation criteria described in the protocol are met.

End of treatment will occur within 7 (+7) days after the SOT201 discontinuation, and Follow-up period.

Every 30 (±2) days until 90 (+7) days after the final dose of SOT201, until disease progression, the start of new anticancer therapy, death, or withdrawal of participant's consent, whichever comes first.

ELIGIBILITY:
Criteria: Inclusion criteria:

Type of patients

* Patients with histologically or cytologically confirmed advanced or metastatic solid tumors who have disease progression after treatment with available therapies for their disease that are known to confer clinical benefit
* Have measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology; lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Accessible tumor tissue available for fresh biopsy or being considered for tumor biopsy according to the treating institution's guidelines and willing to undergo a new biopsy if not clinically contraindicated Note: Newly obtained tumor tissue (to be taken at baseline) is preferred to an archival sample. All tumor biopsies will be collected from the same target lesion, if possible. Archived, fixed tumor tissue may only be collected (taken ideally after completion of the most recent systemic tumor therapy and within 6 months prior to the first dose of trial treatment) if fresh biopsy at screening cannot be retrieved from patients due to safety concerns.
* Performance status: Eastern Cooperative Oncology Group (ECOG) performance score 0-1
* Must have recovered from all adverse events (AEs) due to previous therapies to grade ≤1 toxicity (excluding alopecia) or have stable grade 2 neuropathy as per investigators judgement Note: grade >1 immune- related AEs to any prior treatments may be accepted if considered clinically nonsignificant and/or clinically stable on supportive therapy.
* Organ function: Have adequate organ function during screening and prior to first SOT201 dose.

Exclusion criteria:

Prior/concomitant therapy

* Known clinically relevant intolerability or severe hypersensitivity to prior anti PD-1 or anti-PD-L1 agent therapy, pembrolizumab and/or any of its excipients, or an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, CD134 [OX40], CD137) that caused permanent discontinuation of the agent, or that were grade 4 in severity or have not resolved to grade ≤1.
* Prior exposure to drugs that are agonists or antagonists of IL-2, IL-4, IL-7, IL-8, IL-9, IL-12, IL-15, IL-18, IL-21 or IL-27 prior to ICF signature.
* Prior systemic anti-cancer therapies, including investigational agents, prior to day 1 cycle 1 signature if not otherwise indicated:

  * Less than 3 weeks for all systemic chemotherapy
  * Less than 3 weeks or 5 half-lives (whichever shorter) for any biologic agents
  * Less than 4 weeks for ICIs (targeting CTLA-4, or PD-L1, including e.g., ipilimumab, atezolizumab, avelumab, durvalumab, cemiplimab) prior to cycle 1 day 1
  * Less than 4 weeks from major surgeries and not recovered adequately from the procedure and/or any complications from the surgery before starting SOT201
* Has received radiation therapy ≤14 days before day 1 of cycle 1 or has not recovered to grade ≤1 from treatment-related side effects. A 1-week radiation-free period is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system disease.
* Use of prohibited medication prior or during the course of the trial as specified in the protocol
* Predicted life expectancy ≤3 months
* Clinically significant cardiac abnormalities
* Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years (patients who have had a transplant more than 5 years ago are eligible as long as there are no symptoms of graft versus host disease)
* Diagnosis of other forms of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of SOT201
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years. Patients with basal cell carcinoma of the skin or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known active central nervous system metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during trial screening), clinically stable and without requirement of steroid treatment for at least 14 days before the first dose of SOT201.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy, except in cases for treatment of HIV and/or Hepatitis B
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator

NOTE: Other Inclusion/Exclusion criteria may apply. The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number and percentages of participants with treatment-emergent adverse events (TEAEs) | from patient signing the ICF up to 90 (+7) days after the last dose of SOT201, assessed approximately up to 3 years
  A TEAE is defined as an AE that started or worsened at or after the start of trial treatment Presence of TEAEs, SAEs, and lab abnormalities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Number of participants with dose-limiting toxicities (DLTs) | 21 days of Cycle 1 plus 7 days of cycle 2 per cycle
  DLTs will be defined using NCI CTCAE version 5.0

SECONDARY OUTCOMES:
Characterization of area under the curve (AUClast, AUCinf, AUCtau) of SOT201 | From Day 1 Cycle 1 to Cycle 3, from cycle 4 every other cycle (4, 6, 8), and from cycle 8 at quarterly frequency (11, 14, 17.) until cycle 20
  Area under the concentration versus time curve calculated using the trapezoidal method during a dosing interval (tau)
Characterization of maximum concentration (Cmax) of SOT201 | Time Frame: From Day 1 of Cycle 1 to Cycle 3, from cycle 4 every other cycle (4, 6, 8), and from cycle 8 at quarterly frequency (11, 14, 17.) until cycle 20]
  Maximum plasma concentration observed
Characterization of time to maximum concentration (Tmax) of SOT201 | From Day 1 of Cycle 1 to Cycle 3, from cycle 4 every other cycle (4, 6, 8), and from cycle 8 at quarterly frequency (11, 14, 17..) until cycle 20
  Time to maximum concentration of SOT201
Characterization of pre-dose concentration (Ctrough) of SOT201 | From Day 1 of Cycle 1 to Cycle 3, from cycle 4 every other cycle (4, 6, 8), and from cycle 8 at quarterly frequency (11, 14, 17..) until cycle 20
  Pre-dose trough SOT201 concentrations
Objective response rate (ORR) | From Day 1 of Cycle 1 until disease progression or start new anticancer therapy, whichever comes first, assess to up to approximately 3 years
  Proportion of patients who have a confirmed complete response (CR) or a partial response (PR), as the best overall response (BOR) determined by the Investigator as per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Duration of response (iDoR) | From Day 1 of Cycle 1 until disease progression or start new anticancer therapy, whichever comes first, assess to up to approximately 3 years
  DoR is defined as the time from first documented evidence of confirmed CR or PR until progressive disease (PD) determined by Investigator per RECIST 1.1 or death from any cause, whichever occurs first
Clinical benefit rate (iCBR) | From Day 1 of Cycle 1 until disease progression or start new anticancer therapy, whichever comes first, assess to up to approximately 3 years
  including confirmed CR or PR at any time or stable disease (SD) of at least 6 months determined by Investigator per RECIST 1.1
Progression-free survival (iPFS) | From Day 1 of Cycle 1 until disease progression or start new anticancer therapy, whichever comes first, assess to up to approximately 3 years
  PFS is defined as the time from the date of first administration of IMP to the date of the first documented disease progression determined by Investigator as per RECIST 1.1 or death from any cause, whichever occurs first
Incidence of anti-drug antibodies (ADAs) against SOT201 | Day 1 until 30 (±2) days after the last dose of SOT201
  Incidence of patients with anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, FCAP, Principal Investigator — M.D. Anderson Cancer Center
Locations (7):
- MD Anderson Cancer Center, Houston, Texas, United States
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen (UZA), Edegem, Antwerp
  - Institut Jules Bordet, Anderlecht, Brussels Capital
- Czechia (2):
  - Masarykův Onkologický Ústav, Brno
  - Fakultni Nemocnice Olomouc (FNOL) - Onkologicka Klinika, Olomouc
- Institut Gustave Roussy, Paris, France
- Hospital Universitari Vall d'Hebron - Vall d'Hebron Institut d'Oncologia (VHIO), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matuskova H, Marasek P, Mazhara V, Simonova E, Kosinova L, Danek P, Danova K, Sajnerova K, Malatova I, Hrabankova K, Greco D, Martinec O, Fabisik M, Podzimkova N, Hladikova K, Behalova K, Antosova Z, Sirova M, Mikyskova R, Reinis M, Kovar M, Bechard D, Moebius U, Palova Jelinkova L, Spisek R, Steegmaier M, Adkins I. Novel PD-1-targeted, activity-optimized IL-15 mutein SOT201 acting in cis provides antitumor activity superior to PD1-IL2v. J Immunother Cancer. 2025 Apr 17;13(4):e010736. doi: 10.1136/jitc-2024-010736. PMID 40250867